CLINICAL TRIAL: NCT00026221
Title: A Phase 2 Study of Bevacizumab and Interferon-Alpha-2b in Metastatic Malignant Melanoma
Brief Title: Bevacizumab With or Without Interferon Alfa in Treating Patients With Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00006; NCI-2009-00006 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000069010; 2001C0185; OSU-01H0185; 0132; NCI-2669; OSU 0132 (Other: Ohio State University Comprehensive Cancer Center); 2669 (Other: CTEP); N01CM62207 (NIH); R21CA093071 (NIH); P30CA016058 (NIH)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Recurrent Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — Interferon-alpha; Bevacizumab

ARMS (3):
- Arm I (monoclonal antibody and biological therapy) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive low-dose interferon alfa (IFN-alpha) SC on days 1-14.
  Interventions: Biological: Recombinant Interferon Alfa; Biological: Bevacizumab
- Arm II (monoclonal antibody) (Experimental): Patients receive bevacizumab as in arm I.
  Interventions: Biological: Bevacizumab
- Arm III (monoclonal antibody and biological therapy) (Experimental): Patients receive bevacizumab as in arm I. Patients also receive high-dose IFN-alpha SC on days 1, 3, 5, 8, 10, and 12.
  Interventions: Biological: Recombinant Interferon Alfa; Biological: Bevacizumab

INTERVENTIONS:
Biological: Recombinant Interferon Alfa — Given SC
  Other Names: IFN-A
  Arms: Arm I (monoclonal antibody and biological therapy); Arm III (monoclonal antibody and biological therapy)
Biological: Bevacizumab — Given IV
  Other Names: Avastin; rhuMab-VEGF

SUMMARY:
This randomized phase II trial is studying giving bevacizumab together with interferon alpha to see how well it works compared to giving bevacizumab alone in treating patients with metastatic malignant melanoma. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or deliver cancer-killing substances to them. Interferon alpha may interfere with the growth of the cancer cells and slow the growth of the tumor. Combining bevacizumab with interferon alpha may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the objective response rate and progression-free survival in patients with metastatic malignant melanoma treated with bevacizumab with or without low- or high-dose interferon alpha.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive bevacizumab intravenously (IV) over 30-90 minutes on day 1. Patients also receive low-dose interferon alpha (IFN-alpha) subcutaneously (SC) on days 1-14.

ARM II: Patients receive bevacizumab as in arm I.

ARM III: Patients receive bevacizumab as in arm I. Patients also receive high-dose IFN-alpha SC on days 1, 3, 5, 8, 10, and 12. In all arms, treatment repeats every 14 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients undergo restaging at the completion of course 12. Patients with stable disease or a clinical response may continue treatment according to their assigned treatment arm for up to 1 year. Patients with stable disease after 1 year of treatment with bevacizumab and IFN-alpha (arms I and III) may continue to receive bevacizumab alone every 21 days (as in arm II) in the absence of disease progression.

Patients are followed every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed cutaneous malignant melanoma

  * Must meet one of the following criteria:

    * Clinical evidence of metastatic disease
    * Unresectable regional lymphatic disease
    * Extensive in transit recurrent disease
* Measurable disease

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral computed tomography (CT) scan
* No known brain metastases
* No ocular melanoma
* Performance status - Eastern Cooperative Oncology Group (ECOG) 0-2
* Performance status - Karnofsky 60-100%
* More than 6 months
* White blood cells (WBC) at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No clinical evidence of coagulopathy
* Bilirubin =< 2.0 mg/dL (3.0 mg/dL for patients with Gilbert's disease provided patient is stable and asymptomatic)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) no greater than 2.5 times upper limit of normal (ULN)
* Prothrombin time (PT)/International normalized ratio (INR) less than 1.5
* Creatinine =< 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* Protein < 1,000 mg on 24-hour urine collection for patients with proteinuria >= 1+
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No history of thrombosis (e.g., deep vein thrombosis), unless the following criteria are met:

  * INR in normal range (usually 2-3) AND on a stable dose of warfarin or low molecular weight heparin
  * No active bleeding or pathologic condition that would confer a high risk of bleeding (e.g., known varices or tumor involving major vessels)
* No uncontrolled hypertension
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reactions to compounds of similar chemical or biologic composition to bevacizumab or interferon alfa
* No ongoing or active infection
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* Human immunodeficiency virus (HIV) allowed provided otherwise well
* At least 4 weeks since prior adjuvant interferon alfa
* No prior interferon alfa for metastatic disease
* No prior cytokine therapy for metastatic disease (e.g., high-dose interleukin-2 [IL-2])

  * Prior IL-2 allowed for patients randomized to arm III only
* No prior investigational antiangiogenic agents
* No more than 1 prior chemotherapy regimen for metastatic disease
* At least 4 weeks since prior chemotherapy and recovered
* At least 4 weeks since prior radiotherapy and recovered
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2001-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Carson, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Bevacizumab + Iinterferon-alpha-2b: Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive low-dose interferon alfa (IFN-alpha) SC on days 1-14.
  Recombinant Interferon Alfa: Given SC
  Bevacizumab: Given IV
- Arm II: Bevacizumab Alone: Patients receive bevacizumab as in arm I.
  Bevacizumab: Given IV
Period: Overall Study
Arm/Group | Arm I: Bevacizumab + Iinterferon-alpha-2b | Arm II: Bevacizumab Alone | Arm III (Monoclonal Antibody and Biological Therapy)
Started | 16 | 16 | 25
Completed | 16 | 16 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Monoclonal Antibody and Biological Therapy) | Arm II (Monoclonal Antibody) | Arm III (Monoclonal Antibody and Biological Therapy) | Total
Number analyzed (Participants) | 16 | 16 | 25 | 57
Age, Continuous [Median (Full Range); unit: years] | 64 [28 to 74] | 54 [39 to 83] | 58.4 [31 to 79] | 57 [28 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 9 | 23
  Male | 9 | 9 | 16 | 34
Region of Enrollment [Number; unit: patients]
  United States | 16 | 16 | 25 | 57

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Measured from the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: Up to 2 years
Measure: Number; unit: patients
Arm/Group | Arm I: Bevacizumab + Iinterferon-alpha-2b | Arm II: Bevacizumab Alone | Arm III (Monoclonal Antibody and Biological Therapy)
Number analyzed (Participants) | 15 | 16 | 25
patients | 1 | 0 | 6

2. Other Pre Specified Outcome: Toxicity
Description: Evaluated using the National Cancer Institute (NCI) Common Toxicity Criteria version 2.0.
Time Frame: Continuously from the start of treatment to the end of study
Reporting Status: Not Posted

3. Primary Outcome: Progression-free Survival
Description: Defined as the time from treatment start date until documentation of progressive disease. Evaluated using the new international criteria proposed by the RECIST Committee. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Arm I: Bevacizumab + Iinterferon-alpha-2b | Arm II: Bevacizumab Alone | Arm III (Monoclonal Antibody and Biological Therapy)
Number analyzed (Participants) | 15 | 16 | 25
months | 3 [1.5 to 10] | 8.5 [1 to 47] | 4.8 [.9 to 62.5]

4. Secondary Outcome: Comparison of Plasma Levels of VEGF Following Administration of Bevacizumab Alone or in Combination With IFN-alfa
Description: Analyzed by Enzyme-Linked Immunosorbent Assay (ELISA).VEGF only analyzed at baseline.
Time Frame: At baseline
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Arm I: Bevacizumab + Iinterferon-alpha-2b | Arm II: Bevacizumab Alone | Arm III (Monoclonal Antibody and Biological Therapy)
Number analyzed (Participants) | 16 | 16 | 25
pg/mL | 567 [293 to 9719] | 633 [212 to 9810] | 18 [0 to 412]

5. Secondary Outcome: New Vessel Formation in Patient Tumor Samples
Description: Evaluated using immunohistochemistry.
Time Frame: Up to 2 years
Population: Data were not collected and not assessed.
Arm/Group | Arm I: Bevacizumab + Iinterferon-alpha-2b | Arm II: Bevacizumab Alone | Arm III (Monoclonal Antibody and Biological Therapy)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: The NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3 was utilized for Adverse Event reporting.
Arm/Group | Arm I: Bevacizumab + Iinterferon-alpha-2b | Arm II: Bevacizumab Alone | Arm III (Monoclonal Antibody and Biological Therapy)
Serious Adverse Events (participants affected / at risk) | 1/16 | 2/16 | 3/25
Other Adverse Events (participants affected / at risk) | 5/16 | 16/16 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Bevacizumab + Iinterferon-alpha-2b (N=16) | Arm II: Bevacizumab Alone (N=16) | Arm III (Monoclonal Antibody and Biological Therapy) (N=25)
Subdural Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Elevated Troponin level (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Emboli (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombolembolic event (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I: Bevacizumab + Iinterferon-alpha-2b (N=16) | Arm II: Bevacizumab Alone (N=16) | Arm III (Monoclonal Antibody and Biological Therapy) (N=25)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) — Grade 3
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) — Grade 3
Fatigue (General disorders) | 2 (2) | 3 (3) | 3 (3) — Grade 3
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) — Grade 3
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) — Grade 3
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 0 (0) — Grade 3
Mental Status Changes (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — Grade 3
Pain (General disorders) | 5 (5) | 4 (4) | 0 (0) — Grade 3
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 3 (3) — Grade 3
Thrombosis/embolism (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) — Grade 3 and 4
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) — Grade 3 and 4
Confusion/Memory loss (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) — Grade 3 and 4
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) — Grade 3 and 4
Neutropenia (General disorders) | 0 (0) | 0 (0) | 5 (5) — Grade 3 or 4
AST/ALT (Investigations) | 0 (0) | 0 (0) | 2 (2) — Grade 3 and 4
Abdominal pain/cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) — Grade 3 and 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less